CLINICAL TRIAL: NCT01977898
Title: Incidence of Post-Dural Puncture Headache Following Unintentional Dural Puncture: A Randomized Trial of Intrathecal Morphine Versus Saline
Brief Title: Incidence of Headache Following an Unintentional Dural Puncture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Feyce M. Peralta, MD, MS, Assistant Professor in Anesthesiology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU00043549
Record Dates: First submitted 2013-10-31; First posted 2013-11-07 (Estimated); Results first posted 2021-04-02 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Postdural Puncture Headache; Post-Lumbar Puncture Headache; Cerebrospinal Fluid Leaks
Keywords: Postdural puncture headache; Intrathecal morphine; Intrathecal catheter; Headache; Labor and delivery; Unintentional dural puncture
MeSH Terms: conditions — Post-Dural Puncture Headache; Cerebrospinal Fluid Leak; Headache | interventions — Morphine; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Morphine (Experimental): Patients randomized to the treatment group (morphine) will receive preservative-free morphine 0.3 mL (150 mcg) intrathecally.
  Interventions: Drug: Morphine
- Saline (Placebo Comparator): Patients randomized to the control group will receive normal saline 0.3 mL intrathecally.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Morphine — The drug will be prepared in tuberculin syringes. After thoroughly sanitizing the catheter port with a Chloroprep wipe and allowing adequate time for drying of the Chloroprep, the anesthesiologist will first attach a 3-mL syringe to the catheter port and aspirate to a volume of 1 mL. This syringe will then be removed from the port. The study drug will then be administered through the intrathecal catheter via the tuberculin syringe. The 3-mL syringe containing the aspirate will then be injected via the catheter, effectively flushing the study drug through the catheter. The intrathecal catheter will be removed immediately following the injection.
  Other Names: Duramorph
  Arms: Morphine
Drug: Saline — The drug will be prepared in tuberculin syringes. After thoroughly sanitizing the catheter port with a Chloroprep wipe and allowing adequate time for drying of the Chloroprep, the anesthesiologist will first attach a 3-mL syringe to the catheter port and aspirate to a volume of 1 mL. This syringe will then be removed from the port. The study drug will then be administered through the intrathecal catheter via the tuberculin syringe. The 3-mL syringe containing the aspirate will then be injected via the catheter, effectively flushing the study drug through the catheter. The intrathecal catheter will be removed immediately following the injection.
  Other Names: Normal Saline
  Arms: Saline

SUMMARY:
The purpose of this study is to evaluate the use of intrathecal morphine administration following an unintentional dural puncture, to decrease the incidence of post dural puncture headaches (PDPH) in obstetric patients.

DETAILED DESCRIPTION:
Unintentional dural puncture is a known risk of neuraxial techniques, occurring in roughly 1% of all epidural catheter placements. The incidence of post dural puncture headaches(PDPH) after unintentional dural puncture (UDP) is 50-80%. A PDPH is defined as a headache that occurs following a dural puncture, worsens within 15 minutes after sitting or standing and improves within 15 minutes after lying, with at least one of the following: neck stiffness, tinnitus, hypacusia, photophobia, or nausea. The headache develops within 5 days after dural puncture and resolves either spontaneously within 1 week or within 48 hours after effective treatment of the spinal fluid leak.

The rates of PDPH following unintentional dural puncture with placement of an intrathecal catheter will be compared in two groups: intrathecal morphine (treatment) versus intrathecal saline (control) administered 1-2 hours after delivery, followed by immediate catheter removal. Patients randomized to the treatment group (morphine) will receive preservative-free morphine 0.3 mL (150 mcg) intrathecally. Those randomized to the control group will receive normal saline 0.3 mL intrathecally. After administration of intrathecal morphine, all patients will have their respirations monitored every hour for a period of 12 hours and then every two hours for a period of 12 hours. On postpartum days 1-5, all patients will be visited daily while inpatient and/or contacted by phone after discharge from the hospital.

PDPH can lead to significant morbidity and negatively impact patient satisfaction with postpartum recovery. Along with headache, patients may develop cranial nerve palsy during the postpartum period leading to permanent disability. In addition, new mothers are unable to bond with their babies due to headache and associated symptoms of nausea, vomiting and limited mobility secondary to pain. Therefore, an effective intervention to decrease the risk of PDPH after UDP would be useful.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum patients following vaginal delivery
* Unintentional dural puncture
* Functioning intrathecal catheter
* Patients must be 18 years of age or older
* English speaking.

Exclusion Criteria:

* History of previous PDPH
* Body mass index BMI > 40 kg/m2
* History of obstructive sleep apnea (OSA)
* Morphine allergy
* Patients who receive Cesarean delivery

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2011-11; Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Feyce Peralta, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Apfel CC, Saxena A, Cakmakkaya OS, Gaiser R, George E, Radke O. Prevention of postdural puncture headache after accidental dural puncture: a quantitative systematic review. Br J Anaesth. 2010 Sep;105(3):255-63. doi: 10.1093/bja/aeq191. Epub 2010 Aug 3. PMID 20682567
- [Background] Denny N, Masters R, Pearson D, Read J, Sihota M, Selander D. Postdural puncture headache after continuous spinal anesthesia. Anesth Analg. 1987 Aug;66(8):791-4. No abstract available. PMID 3605700
- [Background] Choi PT, Galinski SE, Takeuchi L, Lucas S, Tamayo C, Jadad AR. PDPH is a common complication of neuraxial blockade in parturients: a meta-analysis of obstetrical studies. Can J Anaesth. 2003 May;50(5):460-9. doi: 10.1007/BF03021057. PMID 12734154
- [Background] Choi A, Laurito CE, Cunningham FE. Pharmacologic management of postdural puncture headache. Ann Pharmacother. 1996 Jul-Aug;30(7-8):831-9. doi: 10.1177/106002809603000722. PMID 8826568
- [Background] Hartopp R, Hamlyn L, Stocks G. Ten years of experience with accidental dural puncture and post-dural-puncture headache in a tertiary obstetric anaesthesia department. Int J Obstet Anesth. 2010 Jan;19(1):118. doi: 10.1016/j.ijoa.2009.06.004. Epub 2009 Nov 28. No abstract available. PMID 19945855
- [Background] Angle P, Tang SL, Thompson D, Szalai JP. Expectant management of postdural puncture headache increases hospital length of stay and emergency room visits. Can J Anaesth. 2005 Apr;52(4):397-402. doi: 10.1007/BF03016283. PMID 15814755
- [Background] Carbaat PA, van Crevel H. Lumbar puncture headache: controlled study on the preventive effect of 24 hours' bed rest. Lancet. 1981 Nov 21;2(8256):1133-5. doi: 10.1016/s0140-6736(81)90586-9. No abstract available. PMID 6118577
- [Background] Sudlow C, Warlow C. Posture and fluids for preventing post-dural puncture headache. Cochrane Database Syst Rev. 2002;(2):CD001790. doi: 10.1002/14651858.CD001790. PMID 12076420
- [Background] Hakim SM. Cosyntropin for prophylaxis against postdural puncture headache after accidental dural puncture. Anesthesiology. 2010 Aug;113(2):413-20. doi: 10.1097/ALN.0b013e3181dfd424. PMID 20613476
- [Background] Carter BL, Pasupuleti R. Use of intravenous cosyntropin in the treatment of postdural puncture headache. Anesthesiology. 2000 Jan;92(1):272-4. doi: 10.1097/00000542-200001000-00043. No abstract available. PMID 10638928
- [Background] Ayad S, Demian Y, Narouze SN, Tetzlaff JE. Subarachnoid catheter placement after wet tap for analgesia in labor: influence on the risk of headache in obstetric patients. Reg Anesth Pain Med. 2003 Nov-Dec;28(6):512-5. doi: 10.1016/s1098-7339(03)00393-6. PMID 14634940
- [Background] Charsley MM, Abram SE. The injection of intrathecal normal saline reduces the severity of postdural puncture headache. Reg Anesth Pain Med. 2001 Jul-Aug;26(4):301-5. doi: 10.1053/rapm.2001.22584. PMID 11464346
- [Background] Cohen S, Amar D, Pantuck EJ, Singer N, Divon M. Decreased incidence of headache after accidental dural puncture in caesarean delivery patients receiving continuous postoperative intrathecal analgesia. Acta Anaesthesiol Scand. 1994 Oct;38(7):716-8. doi: 10.1111/j.1399-6576.1994.tb03983.x. PMID 7839783
- [Background] Scavone BM, Wong CA, Sullivan JT, Yaghmour E, Sherwani SS, McCarthy RJ. Efficacy of a prophylactic epidural blood patch in preventing post dural puncture headache in parturients after inadvertent dural puncture. Anesthesiology. 2004 Dec;101(6):1422-7. doi: 10.1097/00000542-200412000-00024. PMID 15564951
- [Background] Eldor J, Gozal Y, Lavie A, Guedj P. Late postspinal headache treated with epidural morphine. Anaesthesia. 1990 Dec;45(12):1099. doi: 10.1111/j.1365-2044.1990.tb14936.x. No abstract available. PMID 2278354
- [Background] Al-metwalli RR. Epidural morphine injections for prevention of post dural puncture headache. Anaesthesia. 2008 Aug;63(8):847-50. doi: 10.1111/j.1365-2044.2008.05494.x. Epub 2008 Jun 10. PMID 18547293
- [Background] Banks S, Paech M, Gurrin L. An audit of epidural blood patch after accidental dural puncture with a Tuohy needle in obstetric patients. Int J Obstet Anesth. 2001 Jul;10(3):172-6. doi: 10.1054/ijoa.2000.0826. PMID 15321606
- [Background] Olesen J, Steiner TJ. The International classification of headache disorders, 2nd edn (ICDH-II). J Neurol Neurosurg Psychiatry. 2004 Jun;75(6):808-11. doi: 10.1136/jnnp.2003.031286. PMID 15145989

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 68 were consented to participate in the study . 2 withdrew and 3 were excluded for non-functional catheter.
Period: Overall Study
Arm/Group | Morphine | Saline
Started | 28 | 35
Completed | 27 | 34
Not Completed | 1 | 1
Not completed — Non functioning catheter | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Morphine | Saline | Total
Number analyzed (Participants) | 27 | 34 | 61
Age, Continuous [Median (Full Range); unit: Years] | 33 [30 to 36] | 32 [29 to 34] | 32 [29 to 36]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 34 | 61
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 5 | 6
  White | 24 | 26 | 50
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 27 | 34 | 61
Ethnicity [Count of Participants; unit: Participants]
  Hispanic (ethnicity) | 7 | 3 | 10
  Non-hispanic (ethnicity) | 20 | 31 | 51
Body Mass Index (kg/m^2) [Median (Inter-Quartile Range); unit: kg/m^2] — Body mass index (BMI) is derived from the (weight) and height of the subject. The BMI is defined as the body mass divided by the square of the body height, and is expressed in units of kg/m^2.
  kg/m^2 | 29.1 [25.3 to 33.0] | 28.9 [25.5 to 33.9] | 29.0 [25.3 to 33.9]
Nulliparous [Count of Participants; unit: Participants] — Number of participants who presented as nulliparous.
  Participants | 5 | 4 | 9
Gestational age (weeks) [Median (Full Range); unit: Weeks] | 39 [38 to 40] | 39 [38 to 40] | 39 [38 to 40]
Loss of resistance method [Count of Participants; unit: Participants] — Loss of resistance method of catheter placement (either air or saline) used by the operator.
  Participants
    Air | 16 | 17 | 33
    Saline | 11 | 17 | 28
Intrathecal catheter depth (cm) [Median (Inter-Quartile Range); unit: Centimeters (cm)] — The final depth of the placement of the catheter in centimeters.
  Centimeters (cm)
    Insertion | 11 [9.5 to 11] | 11 [10 to 12] | 11 [9.5 to 12]
    Removal | 11 [9.5 to 11] | 11 [10 to 12] | 11 [9.5 to 12]
Unable to aspirate prior to administering study drug (n) [Count of Participants; unit: Participants] — The number of subjects whose intrathecal catheter were unable to be aspirated prior to study drug administration.
  Participants | 4 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Participants Who Report Post Dural Puncture Headaches
Description: Participants who report post dural puncture headaches from delivery to postpartum day 5
Time Frame: 5 days
Measure: Count of Participants; unit: Participants
Arm/Group | Morphine | Saline
Number analyzed (Participants) | 27 | 34
Participants | 21 | 27
Statistical Analysis 1: Comparison: Morphine vs Saline; A sample size of 65 patients in each group would be required to achieve 80% power to detect this difference between intrathecal morphine and saline administration . Sample size of 64 per group achieve 80% power to detect a difference between the group proportions of 0.25. The proportion in the treatment group is assumed to be 0.5 under the null hypothesis and 0.25 under the alternative hypothesis. The proportion in the control group is .05.The significance level of the test was targeted at .05; Test type: Superiority; p = .877, Fisher Exact

2. Secondary Outcome: Severity of Post Dural Puncture Headache
Description: Severity of post dural puncture headache on a numerical rating scale 0= no pain and 10= worst pain imaginable from the time of delivery to postpartum day 5.
Time Frame: Time of unintentional dural puncture to postpartum day 5
Population: 21 in the morphine group and 27 in the saline group experienced headaches.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Morphine | Saline
Number analyzed (Participants) | 21 | 27
score on a scale | 7 [3 to 8.5] | 7.5 [5 to 8]
Statistical Analysis 1: Comparison: Morphine vs Saline; Test type: Superiority; p = .499, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Treatment Method for Headache
Description: Treatment method completed for unintentional dural puncture headache.
Time Frame: Unintentional dural puncture - Postpartum day 5
Population: 21 in the morphine group and 27 in the saline group experienced unintentional post dural puncture headaches.
Measure: Count of Participants; unit: Participants
Arm/Group | Morphine | Saline
Number analyzed (Participants) | 21 | 27
Participants
  Epidural blood patch | 11 | 10
  Oral analgesics | 9 | 16
  Hydration | 1 | 1
Statistical Analysis 1: Comparison: Morphine vs Saline; Test type: Superiority; p = .463, Chi-squared

4. Secondary Outcome: Number of Participants With Cranial Nerve Symptoms
Description: The number of participants who experience cranial nerve symptoms up to 5 days after the unintentional dural puncture.
Time Frame: 5 days
Population: 21 in the morphine group and 27 in the saline group experienced unintentional dural puncture headaches.
Measure: Count of Participants; unit: Participants
Arm/Group | Morphine | Saline
Number analyzed (Participants) | 21 | 27
Participants
  None | 13 | 24
  Visual | 1 | 0
  Auditory | 7 | 3
Statistical Analysis 1: Comparison: Morphine vs Saline; Test type: Superiority; p = .0463, Chi-squared

5. Secondary Outcome: Repeat Epidural Blood Patch
Description: Repeated epidural blood patch for headache pain after unintentional dural puncture.
Time Frame: After first epidural blood patch to 5 days after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Morphine | Saline
Number analyzed (Participants) | 11 | 10
Participants | 1 | 1
Statistical Analysis 1: Comparison: Morphine vs Saline; Test type: Superiority; p = .525, Chi-squared

6. Secondary Outcome: Presenting Day of Headache
Description: Presenting day of headache after unintentional dural puncture
Time Frame: Dural puncture to 5 days after delivery
Population: 21 in the morphine group and 27 in the saline group experienced headache after unintentional dural puncture.
Measure: Count of Participants; unit: Participants
Arm/Group | Morphine | Saline
Number analyzed (Participants) | 21 | 27
Participants
  Day 1 | 9 | 11
  Day 2 | 8 | 8
  Day 3 | 1 | 4
  Day 4 | 3 | 4
Statistical Analysis 1: Comparison: Morphine vs Saline; Test type: Superiority; p = 0.691, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Number of Participants With Duration in Days of Headache After Unintentional Dural Puncture.
Description: The duration in days of headaches the participants experience after an unintentional dural puncture
Time Frame: 5 days
Population: 21 in the morphine group and 27 in the saline group experienced headache after unintentional dural puncture.
Measure: Count of Participants; unit: Participants
Arm/Group | Morphine | Saline
Number analyzed (Participants) | 21 | 27
Participants
  1 day | 4 | 8
  2 day | 5 | 9
  3 day | 7 | 4
  4 day | 4 | 5
  5 day | 1 | 1
Statistical Analysis 1: Comparison: Morphine vs Saline; Test type: Superiority; p = 0.610, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Greatest Level of Headache Pain Experienced With the Unintentional Dural Puncture
Description: Greatest reported headache pain associated with unintentional dural puncture reported on a scale of 0= no pain to 10= worst pain imaginable.
Time Frame: 5 days
Population: 21 in the morphine group and 27 in the saline group experienced unintentional post dural puncture headache.
Measure: Median (Full Range); unit: Score on a scale (0=no pain to 10 worst)
Arm/Group | Morphine | Saline
Number analyzed (Participants) | 21 | 27
Score on a scale (0=no pain to 10 worst) | 7 [3 to 8.5] | 7.5 [5 to 8]
Statistical Analysis 1: Comparison: Morphine vs Saline; Test type: Superiority; p = .499, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Intrathecal Catheter Dwell Time
Description: Intrathecal catheter dwell time(time from insertion to time of removal in minutes).
Time Frame: Insertion time to removal in minutes
Measure: Median (Inter-Quartile Range); unit: Insertion to removal time in minutes
Arm/Group | Morphine | Saline
Number analyzed (Participants) | 27 | 34
Insertion to removal time in minutes | 418 [291 to 550] | 427 [286 to 540]
Statistical Analysis 1: Comparison: Morphine vs Saline; Test type: Superiority; p = .06, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Intrathecal Infusion Volume
Description: Intrathecal infusion volume in milliliters
Time Frame: Time of insertion of catheter to time catheter removed
Measure: Median (Inter-Quartile Range); unit: Milliters
Arm/Group | Morphine | Saline
Number analyzed (Participants) | 27 | 34
Milliters | 12.9 [8 to 19.0] | 16.2 [6.9 to 27]
Statistical Analysis 1: Comparison: Morphine; Test type: Superiority; p = .31, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Mode of Delivery
Description: Mode of delivery of the baby (vaginal delivery or instrumented vaginal delivery)
Time Frame: up to 10 hours after intrathecal catheter placed
Measure: Count of Participants; unit: Participants
Arm/Group | Morphine | Saline
Number analyzed (Participants) | 27 | 34
Participants
  Vaginal Delivery | 24 | 29
  Instrumented Vaginal Delivery | 3 | 5

ADVERSE EVENTS:
Time Frame: 5 days after delivery of baby.
Arm/Group | Morphine | Saline
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/34
Other Adverse Events (participants affected / at risk) | 0/27 | 0/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Morphine (N=27) | Saline (N=34)
New onset nausea (Gastrointestinal disorders) | 0 (0) | 0 (0)
New onset vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The results of our study should only be interpreted in the context of its limitations. Our sample size is small and we stopped the study prior to meeting our original estimated sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-09): https://cdn.clinicaltrials.gov/large-docs/98/NCT01977898/Prot_SAP_000.pdf